CLINICAL TRIAL: NCT00716651
Title: A Phase II, Single Center Open Label, Prospective Trial to Evaluate the Efficacy and Safety of Mepolizumab for Patients With Refractory or Relapsing Churg Strauss Syndrome
Brief Title: Safety and Efficacy Study of Mepolizumab in Churg Strauss Syndrome
Acronym: MEPOCHUSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Moosig, PD Dr. Frank Moosig, University Hospital Schleswig-Holstein
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBB1; EudraCT 2006-001791-20
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Churg Strauss Syndrome
MeSH Terms: conditions — Churg-Strauss Syndrome | interventions — mepolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: mepolizumab — 750 mg mepolizumab iv q4wk until week 32

SUMMARY:
Churg-Strauss syndrome is a rare type of systemic vasculitis which occurs almost exclusively in patients with asthma and which is characterized by prominent blood and tissue eosinophilia. The disease has a chronic smoldering course with a permanent need for medium to high corticosteroid doses. Available unselective immunosuppressive agents are often insufficient to reduce corticosteroid doses, to induce complete remission and to protect patients from disease flares which occur in more than 50 % of cases.

Interleukin-5 is the most potent cytokine regulating the production of eosinophil granulocytes which are the major effector cells in Churg-Strauss syndrome. Recently, an increased production of interleukin-5 was demonstrated in Churg-Strauss syndrome. Mepolizumab is a monoclonal IgG antibody targeting interleukin-5 and is effective in the treatment of the HES. The hypothesis of this study is, that mepolizumab will induce remission and allow for steroid reduction.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* documented history of Churg Strauss Syndrome
* active disease
* subjects must complete screening and baseline assessment
* stable corticosteroid dose of > 12.5 mg prednisolone for at least one week
* treatment with cyclophosphamide (pulse or daily oral) or methotrexate or azathioprin or leflunomide in a stable dose for at least 4 weeks
* not pregnant or nursing
* negative pregnancy test and agree to practice birth control

Exclusion Criteria:

* life threatening disease or other critical illness deemed inappropriate for inclusion in the study by the principal investigator
* treatment with other immunosuppressive agents within 4 weeks prior to randomisation
* corticosteroid pulse of > 60 mg within the last three weeks prior to randomisation
* known secondary cause of eosinophilia
* no history or clinical features of vasculitis
* diagnosis of other primary systemic vasculitis
* currently active malignant disease
* abnormal laboratory values
* impaired cardiac function
* history of allergic reaction due to monoclonal antibodies
* prior treatment with anti-hIL-5 monoclonal antibody
* exposure to investigational drug within 30 days prior to randomisation
* positive pregnancy test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-07; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Primary endpoint is the percentage of patients with Churg-Strauss Syndrome that attain remission | 52 weeks

SECONDARY OUTCOMES:
Change in BVAS score | 52 weeks
Change in Disease Extent Index score | 52 weeks
Permanent End organ damage assessed by the Vasculitis Damage Index | 52 weeks
Time to remission | 52 weeks
Response, defined as a 50 % reduction of the BVAS score | 52 weeks
Time to response | 52 weeks
The frequency of relapses | 52 weeks
Blood eosinophil count | 52 weeks
Frequency of all AEs and SAEs | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Schleswig Holstein, Rheumaklinik Bad Bramstetd, Bad Bramstedt, Schleswig-Holstein, Germany